CLINICAL TRIAL: NCT00132119
Title: A Randomized, Double-Blind, Placebo-Controlled, Multi-Center Study to Assess the Efficacy and Safety of Nalmefene HCl in the Treatment of Pathological Gambling
Brief Title: Nalmefene Gambling Study: Study of Nalmefene HCl in the Treatment of Pathological Gambling
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Somaxon Pharmaceuticals (Industry)
Responsible Party: Somaxon Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SP-N0406
Record Dates: First submitted 2005-08-17; First posted 2005-08-19 (Estimated); Last update posted 2008-05-19 (Estimated); Status verified 2008-05

CONDITIONS: Pathological Gambling
MeSH Terms: conditions — Gambling | interventions — nalmefene

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Nalmefene HCl 20 mg
  Interventions: Drug: nalmefene HCl
- 2 (Experimental): Nalmefene HCl 40 mg
  Interventions: Drug: nalmefene HCl
- 3 (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: nalmefene HCl — Nalmefene HCl film-coated tablets, 20 or 40 mg, administered orally once daily for 10 weeks.
  Arms: 1; 2
Other: Placebo — Placebo tablet
  Arms: 3

SUMMARY:
The purpose of this study is to determine if nalmefene is safe and effective in the treatment of pathological gambling.

DETAILED DESCRIPTION:
Randomized, double-blind, placebo-controlled, parallel-group, multi-centered, outpatient study to assess the efficacy, safety and tolerability of two doses of nalmefene in patients with current diagnosis of pathological gambling.

ELIGIBILITY:
Inclusion Criteria:

* Current diagnosis of pathological gambling as defined by Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition, Text Revision (DSM-IV-TR)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 233 (Actual)
Dates: Start 2005-08; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
Assess efficacy in treatment of pathological gambling

SECONDARY OUTCOMES:
Evaluate safety and tolerability in treatment of pathological gambling

CONTACTS AND LOCATIONS:
Overall Officials: Philip Jochelson, MD, Study Director — Somaxon Pharmaceuticals CMO